CLINICAL TRIAL: NCT02438020
Title: Double-blind Randomized Trial Using Oral Metformin Versus Placebo in the Treatment of Acanthosis Nigricans in Children With Obesity
Brief Title: Study of Efficacy of Metformin in the Treatment of Acanthosis Nigricans in Children With Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Juan Pablo Castanedo-Cazares (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Sponsor-Investigator, Juan Pablo Castanedo-Cazares, Dermatology research director, Universidad Autonoma de San Luis Potosí
Organization: Universidad Autonoma de San Luis Potosí (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MET-AN
Record Dates: First submitted 2015-05-03; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Acanthosis Nigricans
Keywords: Acanthosis nigricans; obesity; children; metformin
MeSH Terms: conditions — Acanthosis Nigricans; Obesity | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): 500 mg metformin oral intake before main meal
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo tablet before main meal.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — One tablet of 500 mg will be ingested before the main meal
  Other Names: Glucophage; Glumetza; Fortamet; Riomet
  Arms: Metformin
Other: Placebo — A placebo tablet will be ingested daily before main meal.
  Arms: Placebo

SUMMARY:
Obesity is often accompanied by insulin resistance and/or hyperinsulinemia. Acanthosis nigricans (AN) is a skin condition commonly present on the neck of obese children. Metformin is a useful drug for conditions characterized by insulin resistance.The aim of this study is to compare the efficacy of metformin versus placebo on AN lesions of the neck as well as their effects on metabolic and anthropometric variables in a sample of obese children. This is a 12-week randomized, double-blind randomized trial involving obese children with AN to receive either metformin or placebo.

Evaluations will be performed every three weeks. Clinical, histological and colorimetric assessments of AN lesions will be compared initially and at the conclusion of the study.

DETAILED DESCRIPTION:
Acanthosis nigricans (AN) are lesions affecting localized areas of the skin in persons with obesity and/or hyperinsulinemia. Roughening of the skin is related with histological papillomatosis and the skin darkening is due to hyperkeratosis. Biochemical mechanisms for developing this hyperplastic lesion involve local cutaneous growth factors. Nearly 40% of Native American teenagers have acanthosis nigricans, whereas about 13% of African American, 6% of Hispanic, and less than 1% of white, non-Hispanic children aged 10-19 have clinically apparent acanthosis nigricans. AN is a clinical surrogate of laboratory-documented hyperinsulinemia.

The aim of this study is to compare the efficacy of metformin versus placebo on AN lesions of the neck as well as their effects on metabolic (HOMA, triglycerides, cholesterol) and anthropometric variables (BMI, waist) in a sample of obese children. This is a 12-week randomized, double-blind randomized trial involving obese children with AN to receive either metformin or placebo.

Evaluations will be performed every three weeks. Clinical, histological and colorimetric assessments of AN lesions will be compared initially and at the conclusion of the study. Burke´s scale, papillomatosis and hyperkeratosis, and the L* axis of will be used to measure the AN improvement.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from children and parents.
* Children younger than 18 years.
* Clinical diagnosis of acanthosis nigricans.
* Obesity.

Exclusion Criteria:

* Diabetes mellitus.
* Neurological diseases.
* Congenital diseases.
* Oral treatment for obesity in the last two months.
* Topical treatment for the last two months.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement of acanthosis nigricans | baseline and 12 weeks
  Initial and after intervention assessment of acanthosis nigricans using the quantitative scale of Burke (Diabetes Care 22:1655-1659, 1999).
  Five anatomical sites were chosen to assess the presence and extent of AN: neck, axilla, knuckles, elbows, and knees. The neck and axilla are graded for severity on a scale from 0 to 4. For AN present on the neck, texture of the affected area is also measured on a scale from 0 to 3. Knuckles, elbows, and knees are graded as AN present (1) or absent (0). Score goes from 0 to 14.

SECONDARY OUTCOMES:
Histological improvement of acanthosis nigricans | baseline and 12 weeks
  Epidermal and stratum corneum thickness of 3 mm skin samples obtained from neck will be measured using an image processing software initially and at the end of trial.
Depigmentation of acanthosis nigricans | baseline and 12 weeks
  Quantification of pigmentation change of lesions by means of the L axis of the CIE system. 0 is pure white, 100 y total dark. Initially, and at the end of study.

OTHER OUTCOMES:
Serum fasting insulin | baseline and 12 weeks
  Quantification of serum fasting insulin in pmol/L or mIU/L, at baseline and at the end of the study.
Serum fasting glucose | baseline and 12 weeks
  Quantification of serum fasting glucose in mg/dL.
Serum fasting lipids | baseline and 12 weeks
  Quantification of serum fasting lipids in mg/dL. Cholesterol (HDL, LDL, VLDL) and triglycerides.
Waist measurement | baseline and 12 weeks
  Waist measurement in centimeters.
Quantification of Body mass index (BMI) | baseline and 12 weeks
  BMI It is the measure of body fat based on height and weight. The BMI is the body mass divided by the square of the body height, and expressed in units of kg/m2, resulting from weight in kilograms and height in metres

CONTACTS AND LOCATIONS:
Overall Officials: Bertha Torres-Alvarez, MD, Study Chair — Hospital Central "Dr. Ignacio Morones Prieto"; Juan P Castanedo-Cazares, MD, Study Director — Hospital Central "Dr. Ignacio Morones Prieto"; Francisco Goldaracena-Orozco, MD, Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central Dr.Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Bellot-Rojas P, Posadas-Sanchez R, Caracas-Portilla N, Zamora-Gonzalez J, Cardoso-Saldana G, Jurado-Santacruz F, Posadas-Romero C. Comparison of metformin versus rosiglitazone in patients with Acanthosis nigricans: a pilot study. J Drugs Dermatol. 2006 Oct;5(9):884-9. PMID 17039655
- [Background] Freemark M, Bursey D. The effects of metformin on body mass index and glucose tolerance in obese adolescents with fasting hyperinsulinemia and a family history of type 2 diabetes. Pediatrics. 2001 Apr;107(4):E55. doi: 10.1542/peds.107.4.e55. PMID 11335776
- [Background] Romo A, Benavides S. Treatment options in insulin resistance obesity-related acanthosis nigricans. Ann Pharmacother. 2008 Jul;42(7):1090-4. doi: 10.1345/aph.1K446. Epub 2008 May 20. PMID 18492785